CLINICAL TRIAL: NCT04588558
Title: Investigation of the Effectiveness of a Structured Squat-based Program in Knee Osteoarthritis Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, hazal genc, Phd(c), Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hazalgenc
Record Dates: First submitted 2020-10-08; First posted 2020-10-19 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis Knees Both; Pain, Chronic; Walking, Difficulty
Keywords: Osteoarthritis, Knee; Muscle Activation; Exercise; Pain; Fly wheel
MeSH Terms: conditions — Chronic Pain; Mobility Limitation; Osteoarthritis, Knee; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Squat based exercise will be applied to the first group with isoinertial system. Electrotherapy (TENS, ultrasound and hot pack or cold pack) and squat-based home exercise program will be applied to the second group, and only squat-based home exercise program will be applied to the third group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flywheel exercise (Experimental): The term isoinertial is derived from the words iso (same) and inertial (resistance), which define the primary concept of the isoinertial system in a terminology or that expresses both the concentric and eccentric phases of the same muscle contraction. Isoinertial refers to resistance used in exercise training, maintaining a constant inertia throughout the range of motion, a constant resistance in all respects, and facilitating maximum muscle strength. All participants received home exercise for 8 weeks.
  Interventions: Device: Flywheel exercise
- Electrotherapy modality (Active Comparator): Electrotherapy modalities especially transcutaneous electrical nerve stimulation (TENS) and ultrasound is used to treat OA.
  All participants received home exercise for 8 weeks.
  Interventions: Device: Electrotherapy group
- Home exercise (Active Comparator): All participants received home exercise three times a week for 8 weeks. Home exercises are structured with squats. The exercise program includes stretching exercises and strengthening (isometric and isotonic) exercises.
  Interventions: Other: Home exercise

INTERVENTIONS:
Device: Flywheel exercise — Flywheel training is a strength training modality that offers the possibility of performing exercises with eccentric overload and variable resistance as compared to conventional gravity-based resistance training. Flywheel exercise applied three days a week for 8 weeks
  Arms: Flywheel exercise
Other: Home exercise — The active ROM exercise was performed via knee in extension to full-flexion, then knee in flexion to full-extension exercises, repeated 10 times. The strengthening exercises consisted of quadriceps strengthening by holding maximal isometric contractions for 10 s and performing 10 repetitions. Stretching targeted the gastrocnemius- soleus and hamstring muscle and was performed by asking the patient to stretch the muscle for 30 s and to complete three repetitions for each muscle group.
  Arms: Home exercise
Device: Electrotherapy group — The participants in the electrotherapy group received TENS (Intellect; Chattanooga Group, Hixson, TN), therapeutic ultrasound (Intellect 340 Combo) and exercise. TENS was applied via four electrodes around the knee joint: two on the medial and two on the lateral aspect on either side of the joint line for approximately 20 min. For pain relief, the devices were set to a continuous mode (110 Hz, 50 μ). Electrical pulses were asymmetric and biphasic.
  Therapeutic pulsed ultrasound therapy was administered using a 1-MHz frequency, 0.8 W/cm power ultrasound device with a sound-head area of 5 cm2 and effective radiating area of 3.5-5 cm2 . Ultrasound was applied to the medial and lateral parts of the knee in circular movements for a duration of 5 min with the patient in a supine position.
  All participants received the same standardized exercise program. The exercises included aerobic, active ROM, strength, and stretching exercises
  Arms: Electrotherapy modality

SUMMARY:
The main purpose of the study is to examine the effect of squat-based exercise approach in individuals with knee osteoarthritis.

The aim of this study is to compare effect to three groups (flywheel exercise group, electrotherapy modality group and home exercise group) and also decrease the pain, increase muscle strength, activation values and increase the functional level of individuals.

Osteoarthritis is the most common rheumatological disease in the world that primarily results in progressive cartilage destruction. Changes occurring as a result of osteoarthritis are the main cause of disability and are most common in the knee joint.

Osteoarthritis; problems such as pain, tenderness, joint stiffness, joint swelling, movement restriction, joint deformities, loss of muscle strength, decreased functional capacity and impaired quality of life are observed. The daily life activities of individuals with knee osteoarthritis are restricted by the problems of walking up and down stairs, getting out of the chair, standing, squatting, walking.

Improving the symptoms of the disease is an important goal of the rehabilitation process of patients with knee osteoarthritis.

In individuals with knee osteoarthritis, joint structure and deformation in cartilage also show loss of strength with muscles. Strengthening exercises have been used in patients with knee osteoarthritis for a long time. Squat exercise is a type of exercise that is widely used as a strengthening exercise.

DETAILED DESCRIPTION:
OA is endemic around the world. About 30.8 million adults in the United States and 300 million people worldwide live with OA. OA is a disease of the entire joint involving structural changes in articular cartilage, subchondral bone, ligaments, capsule, synovial membrane, and periarticular muscles. Clinically, OA is characterized by joint pain, tenderness, limitation of movement, crepitus, effusion and varying degrees of non-systemic inflammation. Pain, stiffness and difficulty in daily life activities due to the negative impact of functional status are among the main symptoms. The knee is the most affected joint.

The aim of this study is to compare effect to three groups (flywheel exercise, electrotherapy modality and home exercise) Flywheel training is a strength training modality that offers the possibility of performing exercises with eccentric overload and variable resistance as compared to conventional gravity-based resistance training.

Electrophysical agents are used by physiotherapists to treat a wide variety of conditions. Electrotherapy modalities especially transcutaneous electrical nerve stimulation (TENS) and ultrasound is used to treat OA

Hypothesis:

* Ho: Three different protocols applied in individuals with knee osteoarthritis have no effect.
* H1-0: It is effective in three different protocols applied in individuals with knee osteoarthritis, but three don't have statistically effect on each other.
* H1-1: Exercise with isoinertial system in individuals with knee osteoarthritis to be more effective than other treatment protocols
* H1-2: Electrotherapy (TENS, ultrasound and hot pack or cold pack) and squat-based home exercise program is more effective than other treatment protocols in individuals with knee osteoarthritis.
* H1-3: Electrotherapy (TENS, ultrasound and hot pack or cold pack) and squat-based home exercise program in individuals with knee osteoarthritis to be more effective than other treatment protocols

Randomization and blinding

After the baseline assessment, the participants were randomized to one of three intervention groups (ratio 1:1:1) using "Research Randomizer," an online randomization web service (https://www.randomizer.org/).

It was planned as a double-blind study without knowing the necessary treatment or experimental condition for both the subject and the researchers.

Sample size

Sample size was determined using an Instat sample size calculator. In the WOMAC sections, the smallest detectable difference and minimal clinically important difference ranged from 0.51 to 1.33 points. This value was used to calculate the sample size (Angst, Aeschlimann, and Stucki, 2001). Investigators included a two sided alpha value of 0.05, a power of 0.9, and a sample size of 21 per group. To allow for dropouts, the sample size was set at 25 per group.

Risk management:

Failure to reach the number of patients, receiving support from other hospitals of the Medipol Hospital Group Unusual increase in the rate of increase of Covid 19 outbreak, (second wave, permanent curfew): Online controlled (tele-rehabilitation) exercises

Research center

Sefaköy Medipol University Hospital Health Practice and Research Center Statistical method (s) to be used

Statistical analysis will be calculated using SPSS for Windows 22 program.

ELIGIBILITY:
Inclusion Criteria:

1. The age range is between 40-65 years old
2. According to ACR criteria, clinically and radiographically, at least one of the knees should be diagnosed with knee OA (within the last 6 months)
3. Having findings consistent with Kellgren-Lawrence grade II-III OA on knee radiography
4. Pain between 2-7 according to the visual analog scale

Exclusion Criteria:

1. Acute OA in the knee
2. Comorbid diseases (advanced osteoporosis, vertigo, neurological diseases, etc.), injuries and surgeries where exercise is contraindicated
3. Use of NSAIDs and similar disease modifying drugs (Diacerein, Glucosamine etc.) in the last month
4. Having exercised regularly in the last 6 months (more than 1 day a week)
5. Having had arthroplasty surgery
6. Intra-articular injection (hyaluronic acid / steroid) application in the last 6 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 10 minutes
  The primary outcome measures included the level of function determined by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) . WOMAC is a specific, valid, reliable criterion for knee osteoarthritis and includes 24 questions under three subheadings: pain, stiffness and physical function. Each question was scored according to the Likert scale as 0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.

SECONDARY OUTCOMES:
EMG-BF | 10 minutes
  EMG-BF (Intelect Advanced Color Combo + EMG, Chattanooga Group, TN, USA) was used to evaluate muscle activation level. The screen scale was used as a visual feedback, as an increased or decreasing signal tone with varying muscle activity as sensory feedback.
  The undermentioned muscles will be evaluated in study, Rectus femoris Vastus lateralis Vastus medialis Biceps femoris Gastrocnemius
Muscle strength | 10 minutes
  A dynamometer was used to evaluate muscle strength. Muscle strength was evaluated in the following muscles, each measurement was made three times and the average was taken.
  M. Iliopsoas M. Gluteus Maximus M. Gluteus Medius M. Quadriceps Femoris Hamstring muscle group M. Gastrosoleus M. Tibialis Anterior
Algometer | 5 minutes
  The instrument that measures sensitivity to pain and gives a numerical value is called an algometer.
  In total, application was made at 4 different points. Medial point of heel - Right Medial point of heel - Left Medial point of knee-Right Medial point of knee-Left Measurements were made three times and averaged.
Visual Analog Scale (VAS) Evaluation | 5 minutes
  Purpose and application of the test: The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically into numericals. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by placing a point or pointing on this line. Rest, activity and night were evaluated in three different time periods
Time up and go test | 20 seconds
  To determine fall risk and measure the progress of balance, sit to stand and walking.The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down.
30 Seconds Sit To Stand Test | 30 Seconds
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test ( 30CST), is for testing leg strength and endurance in older adults.The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.
Step test | 1 minute
  The individual is asked to climb and descend 7 times. The total time is recorded.
goniometer | 10 minutes
  Lower extremity joints and range of motion were evaluated. Hip Flexion Hip Extension Hip Internal Rotation Hip External Rotation Knee Flexion Knee Extension Ankle Plantar Flexion Ankle Dorsi Flexion

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University Sefaköy Research and Application Hospital, Istanbul, Küçükçekmece, Turkey (Türkiye)